CLINICAL TRIAL: NCT04922996
Title: CaDoBio (Calcium Dobesilate Bioavailability): a Bioavailability and Pharmacokinetics Research Project to Measure the Concentrations of Calcium Dobesilate (Doxium®) in the Nasal Mucosal Tissue, Saliva and Blood of Treated Patients
Brief Title: Bioavailability and Pharmacokinetics of Calcium Dobesilate (Doxium®) in the Nasal Mucosal Tissue, Saliva and Blood of Treated Patients
Acronym: CaDoBio
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Julien Salamun, Principal investigator, University Hospital, Geneva
Other Study IDs: 2020-03050
Record Dates: First submitted 2021-06-03; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Biological Availability
Keywords: Calcium dobesilate; Biological Availability; Pharmacokinetics
MeSH Terms: interventions — Calcium Dobesilate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples Saliva samples Nasal mucosa samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ongoing: Patients already on calcium dobesilate treatment
  Interventions: Drug: Calcium Dobesilate
- New: Patients with approved indication for calcium dobesilate treatment but not already on treatment
  Interventions: Drug: Calcium Dobesilate

INTERVENTIONS:
Drug: Calcium Dobesilate — Dosage of calcium dobesilate in different tissues
  Other Names: Biological samples

SUMMARY:
Calcium dobesilate (CaD) has been shown to have potential antiviral effects, mediated via its interaction with the heparansulfate (HS) binding site of the viral SARS-CoV-2 spike protein (direct action), necessary for interation with the ACE-2 receptor on human cells. Preliminary pre-clinical results using viral pseudotyped particles demonstrated that CaD reduces the uptake of SARS-CoV-2 spike protein in cultured endothelial cells by more than 50%.

Moreover, CaD is a well-established vasoactive and angioprotective drug improving endothelial dysfunction with a good tolerability profile. CaD strengthens vessels integrity and improves blood flow by acting on multiple parameters, like cytokines levels and signaling by FGF and VEGF. All these parameters may be dysregulated at some stage of Covid-19 pathological evolution, and acting on these could potentially reduce the progression toward severe disease. Based on these data, we hypothesize that CaD could be used as an early treatment for SARS-CoV-2 positive outpatients.

However, bioavailability data and pharmacokinetics of CaD are not well known, outside of old data on animal models. Being able to show that the drug is present in nasal mucosae and saliva, where the virus is likely to start the infection of the host, would be a first step before studying a possible effect on the disease course on infected patients.

Therefore this project plans to include between 6 and 10 patients, treated with CaD, for whom different nasal, saliva and blood sample will be taken at different timepoints before and after the daily dose of the treatment. Samples will be then analysed to detect and quantify the presence of CaD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated with calcium dobesilate (1000-2000mg/day), at any time on treatment or for whom initiation of treatment has been prescribed, for one of its Swiss indications:

   * Microangiopathies, in particular diabetic retinopathy.
   * Clinical symptoms of chronic venous insufficiency of the legs (pains, cramps, paraesthesia, oedemas, stasis dermatitis), superficial thrombophlebitis in adjuvant treatment.
   * Haemorrhoidal syndrome, post-thrombotic syndrome, microcirculatory disorders of arteriovenous origin.
2. Male or female
3. Aged ≥18 years
4. Subject has provided the appropriate written informed consent. Subject must provide written informed consent before any study-specific procedures are performed

Exclusion Criteria:

1. Known sensitivity to calcium dobesilate
2. Currently suffering from or treated for a nasal condition, e.g., a runny, congested nose, nasal infection, or an oral condition, e.g., oral infection, including suspected SARS-CoV-2 infection
3. Currently treated with a nasal or an oral product, or any treatment with the same active substance as in CaD (e.g., doxiproct, dicynone)
4. Current participation in any other investigational drug study
5. Only for patients already on CaD treatment: treatment with CaD initiated within last 7 days only
6. Only for patients starting CaD treatment: treatment with CaD within last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients already on CaD treatment according to the approved indication of treatment, or patients meeting conditions for CaD treatment
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
CaD presence and concentration in nasal mucosa | Day 0
  Nasal mucosa tissue of calcium dobesilate for patients on treatment as assessed by tandem mass spectrometry in ug/ml
CaD presence and concentration in saliva | Day 0
  Saliva concentrations of calcium dobesilate for patients on treatment as assessed by tandem mass spectrometry in ug/ml

SECONDARY OUTCOMES:
Pharmakokinetic of CaD in plasma for patients on treatment | Day 0 - before the morning dose
  Calcium dobesilate plasma concentrations in ug/ml for patients on treatment
Pharmakokinetic of CaD in plasma for patients on treatment | Day 0 - 4 hours after the morning dose
  Calcium dobesilate plasma concentrations in ug/ml for patients on treatment
Pharmakokinetic of CaD in plasma for patients on treatment | Day 0 - 8 hours after the morning dose
  Calcium dobesilate plasma concentrations in ug/ml for patients on treatment
Pharmakokinetic of CaD in plasma for patients starting treatment | Day 0 - before the morning dose
  Calcium dobesilate plasma concentrations in ug/ml for patients starting treatment
Pharmakokinetic of CaD in plasma for patients starting treatment | Day 0- 4 hours after the morning dose
  Calcium dobesilate plasma concentrations in ug/ml for patients starting treatment
Pharmakokinetic of CaD in plasma for patients starting treatment | Day 0 - 8 hours after the morning dose
  Calcium dobesilate plasma concentrations in ug/ml for patients starting treatment
Pharmakokinetic of CaD in plasma for patients starting treatment | Day 1 - before the morning dose
  Calcium dobesilate plasma concentrations in ug/ml for patients starting treatment
Pharmakokinetic of CaD in plasma for patients starting treatment | Day 1 - 4 hours after the morning dose
  Calcium dobesilate plasma concentrations in ug/ml for patients starting treatment
Pharmakokinetic of CaD in plasma for patients starting treatment | Day 1- 8 hours after the morning dose
  Calcium dobesilate plasma concentrations in ug/ml for patients starting treatment
Pharmakokinetic of CaD in plasma for patients starting treatment | Day 3- before the morning dose
  Calcium dobesilate plasma concentrations in ug/ml for patients starting treatment
Pharmakokinetic of CaD in plasma for patients starting treatment | Day 3 - 4 hours after the morning dose
  Calcium dobesilate plasma concentrations in ug/ml for patients starting treatment
Pharmakokinetic of CaD in plasma for patients starting treatment | Day 3- 8 hours after the morning dose
  Calcium dobesilate plasma concentrations in ug/ml for patients starting treatment
Pharmakokinetic of CaD in plasma for patients starting treatment | Day 7- before the morning dose
  Calcium dobesilate plasma concentrations in ug/ml for patients starting treatment
Pharmakokinetic of CaD in plasma for patients starting treatment | Day 7 - 4 hours after the morning dose
  Calcium dobesilate plasma concentrations in ug/ml for patients starting treatment
Pharmakokinetic of CaD in plasma for patients starting treatment | Day 7- 8 hours after the morning dose
  Calcium dobesilate plasma concentrations in ug/ml for patients starting treatment
Correlation between nasal mucosal tissue and plasma concentration for patients on treatment | Day 0
  Ratio in %
Correlation between oral tissue and plasma concentration for patients on treatment | Day 0
  Ratio in %

CONTACTS AND LOCATIONS:
Locations (1):
- HUG, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Pharmacokinetic data Individual concentrations